CLINICAL TRIAL: NCT05060497
Title: DYNamic Assessment of Multi Organ Level Dysfunction in Patients Recovering From Covid-19
Acronym: DYNAMOCovid-19
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 20050
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples: Full blood count, renal function including eGFR, troponin, brain natriuretic peptide, glycosylated haemoglobin, liver function, ferritin, creatine kinase (CK), clotting and international normalized ratio (INR), TNF-alpha, IL-6 and CRP
  Muscle biopsy: citrate synthetase
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid patients: Participants who were treated in hospital with laboratory diagnosed Covid-19 requiring high flow oxygen, non invasive ventilation or intubation and have now recovered. They will be recruited 5-7 months post discharge from their local hospital Trust
- Healthy control volunteers: Participants who are otherwise healthy, who have not had Covid-19 infection and are age, gender, BMI and ethnicity matched to patients

SUMMARY:
In this study the investigators are hoping to the find out what changes occur within the body of people recovering from Covid-19 at 5-7 months and 11-13 months following discharge from hospital, compared to healthy controls, and whether these changes can help explain why some patients may experience fatigue. Measurements will be taken using state-of-the-art MRI imaging at rest and also during low intensity exercise, to mimic everyday activity. In doing so it is expected that this will inform ways to adapt exercise rehabilitation programmes, making them better suited for Covid-19 survivors.

DETAILED DESCRIPTION:
Purpose and design Covid-19 manifests as a spectrum of multi-organ damage and dysfunction. Skeletal muscle wasting and strength loss from heightened inflammatory burden and hospital immobilisation, together with vascular dysfunction and lung damage, combine to create a profound insult resulting in severe deconditioning and long-lasting functional insufficiencies. Marked physiological deficits likely prevail due to the multi-organ nature of this insult, but clear understanding of breadth and magnitude is lacking.

Whilst susceptible groups exist, patients surviving this critical illness also include those who were previously fit and well, many of younger and working age, but a unifying trait is the inability to mount a dynamic physiological response to simple every-day activities, such as walking. Greater effort to address the multi-organ nature of this lack of physiological resilience is urgently warranted, it is essential to understand the relative regional contribution of the disease to pathophysiology and frailty. Further, understanding the dynamic response across organs will be fundamental in developing optimal interventions to facilitate recovery.

This project will combine state-of-the-art, validated techniques and research expertise in human physiology, MRI/MRS and clinical medicine to provide novel insight of the impact of Covid-19 on physiological resilience at a multi-organ level (here, muscle, heart and brain related to fatigue/physical activity), using exercise as a stressor. This will provide a unique clinically valuable perspective of whole body dysfunction that will underpin global rehabilitative programmes designed to maximise patient recovery and functionality.

The urgent priority to define Covid-19 multi-organ damage and optimise the rehabilitation package underpins the rapidity of this call.

There are other multi-organ MRI projects post Covid-19 (for example coverscan and C-More) which will take cohorts of patients. DYNAMO differs as it has been developed specifically to mechanistically study the cause for the persisting symptoms such as fatigue, atrophy, impaired exercise tolerance, poor vascular and metabolic health, and cognitive impairment and delineate the targets for rehabilitation. Detailed whole-body and organ level metabolic and physiological assessments will be collected using dynamic magnetic resonance imaging (MRI) and MR spectroscopy measures, with exercise as a stressor, only under stress will some deficits become apparent. This is highly novel, and will deliver unprecedented insight into the mechanisms driving persisting symptoms. DYNAMO will complement other projects, and the objectives and detailed physiological phenotyping described in DYNAMO is not covered elsewhere in other funded imaging studies. Moreover, DYNAMO will provide an important evidence-based foundation for optimising future rehabilitation.

Investigators will be recruiting 30 patients who have recovered from Covid-19, 5-7 months from discharge from their local hospital Trust, compared to 10 age, gender, body mass index (BMI) and ethnicity matched healthy control volunteers. Patients will also undergo a set of 6 month follow up visits to see if there is any change in their physiological and metabolic function.

Recruitment Potentially eligible patients, attending the established post Covid-19 outpatient clinic at the Nottingham University Hospitals Trust as part of their follow up care after hospital admission, will be approached by an existing member of their clinical care team (the Chief investigator (CI) forms part of this team). Similarly, there is active follow-up at other nearby acute hospital trusts in the East Midlands, who are collaborating, from where patients can be recruited. Furthermore, collaborations with PHOSP-Covid on this project have been confirmed and participants who have been involved in PHOSP-Covid can be recruited as a Tier 3 study.

Volunteers will be given a Participant Information Sheet to read about this study and will be advised that with their verbal consent, their contact details can be passed onto a research team, who can contact them to discuss the study further and answer any questions they may have. If needed, the usual hospital interpreter and translator services will be available to assist with discussion of the trial, the participant information sheets, and consent forms, but the consent forms and information sheets will not be available printed in other languages. Potential participants will be given at least 48 hours to decide on whether they wish to participate in the study.

Potential participants may also be approached by way of invitation letter sent to them from their Clinician or a member of the research team, inviting them to consider taking part. A Participant Information Sheet will also be included with this letter. Patients identified through their records by the CI who is also their clinician will be contacted by one of the clinical team who will check/confirm they are in receipt of the letter and discuss the study further, answer any queries and see if they are interested in taking part. They can also contact the study team if they are interested in taking part or leave their contact details so a research nurse can then contact them to discuss the study and /or arrange an appointment to come in for a study visit.

Investigators will also approach participants admitted following Covid-19 related hospital admission to the Nottingham University Hospitals trust, though these patients will be required to wait 5-7 months following discharge to commence study participation.

Any patient who decides to take part in the study will be given an appointment for a study visit; at the start of which, a research fellow (medic), fully trained in the study procedures and informed consent will take consent, participants will have the opportunity to speak to a medically trained doctor if they wish.

In order to recruit volunteers who haven't contracted with Covid, investigators will use our study flyer with relevant contact details, and will advertise on Nottingham University Hospitals and University of Nottingham campuses, in local press, in departmental Facebook and Twitter posts and in any departmental mailing/ emailing lists to people who have agreed to be contacted with such information. A summary of the research study will also be provided on the designated website.

It will be explained to all potential participant that entry into the trial is entirely voluntary and that their treatment and care will not be affected by their decision. It will also be explained that they can withdraw at any time but attempts will be made to avoid this occurrence. In the event of their withdrawal it will be explained that their study research data collected so far cannot be erased and investigators will seek consent to use the data in the final analyses where appropriate. It will be possible to link the withdrawn participant to the log and consent form. However, any personal information, such as contact details will be removed appropriately. Participants that are withdrawn from the study will be replaced with new volunteers.

Volunteers will undergo a series of tests including:

* Height, weight, fat and fat free mass (DEXA scan)
* Blood sampling if not already taken within 1 month of study visit, as part of routine clinical care: Full blood count, renal function including glomerular filtration rate (eGFR), troponin, brain natriuretic peptide, glycosylated haemoglobin, liver function, ferritin, creatine kinase (CK), clotting and inr, Tumour necrosis factor-alpha (TNF-alpha), interlocking-6 (IL-6) and C-reactive protein (CRP)
* Step count over 1 week using Sensewear® armband during waking hours
* Hand grip strength (hand held dynamometer) 3 measurements of grip strength using a hand held dynamometer in the dominant hand.
* Questionnaires: Fatigue severity score, quality of life (Short Form (t-36)), mental health (Personal Health Questionnaire/PHQ), frailty (Rockwood Clinical Frailty Scale/CFS) Dyspnoea-12 and Nottingham activities of daily living, and measure of cognitive state (Montreal Cognitive Assessment/ MoCA), MRI safety questionnaire, DEXA screening form
* ECG
* Arterialised blood gas: using retrograde cannulation
* Spirometry to assess basic lung function if not already done as part of routine clinical care within 1 month of study visit
* Short physical performance battery (SPPB)
* Introduction to the supine exercise equipment and familiarisation (Ergospect diagnostic pedal).
* Whole body glucose disposal during oral glucose tolerance test (OGTT). Fat and carbohydrate oxidation rates in fasting state and in response to OGTT using an indirect calorimetry ventilated hood system will be assessed. Collectively assessing metabolic flexibility, and along with body composition and intramuscular lipid content will provide a powerful index of metabolic health.
* Muscle function assessment (Isokinetic dynamometer) N= 3 maximal voluntary isometric contractions of the knee extensors interspersed with 30 seconds recovery. N=20 repeated isokinetic, knee extensor contractions at a constant angular velocity of 180o/s to determine muscle torque development and fatigue (torque loss).
* Motor unit remodelling using intramuscular EMG (iEMG) to study changes in motor unit size and functionality in the quadriceps muscle group during recovery.
* Quadriceps muscle micro-biopsy for mitochondrial content (citrate synthase maximal activity) - excess muscle tissue will be archived to quantify muscle targets of interest depending on findings
* MR measures (cardiac output, cerebral blood flow and perfusion, oxygen extraction, brain architecture, whole body fat and muscle content and skeletal muscle quality). Measures of cardiac output and structure, brain architecture (grey matter volume and cortical thickness), cerebral blood flow, perfusion, brain fractional oxygen extraction and whole-body fat and muscle volumes will be determined in the resting state. Subjects will then perform a period of steady-state low intensity supine exercise using an in-magnet exercise stepper ergometer (Ergospect diagnostic pedal), during which measures of cardiovascular and cerebrovascular physiological resilience to exercise (ability to respond) will be collected (cardiac output, left ventricular dysfunction, tagging, cerebral blood flow, perfusion and oxygenation).
* Skeletal muscle quality will be assessed using 31P magnetic resonance spectroscopy (31P MRS) of calf muscle Phosphocreatine (PCr) recovery kinetics following within-scanner plantar flexion exercises, using a MRI compatible ergometer (Trispect diagnostic pedal) and muscle proton MRS will be used to quantify intra/extra myocellular lipid content.

ELIGIBILITY:
Inclusion Criteria:

Covid patients -

* Adults aged 18 years and over,
* Severe, laboratory confirmed Covid-19 infection that required hospital admission,
* 5-7 months post discharge from local hospital Trusts.

Controls -

* No active or previous Covid infection, ie no previous positive Covid PCR test and absence of active symptoms
* Matched for age, gender, BMI and ethnicity.

Exclusion Criteria:

* Absolute contraindications for MR scan
* Pre-Covid diagnosed chronic respiratory, renal, cardiovascular or cerebrovascular disease or diabetes
* BMI<20kg/m2
* Pregnancy
* Those requiring oxygen therapy or non-invasive ventilation
* Those on anticoagulation will be included but will not have a muscle biopsy
* Active arthritis
* Overt muscle damage, e.g. plasma creatine kinase > 300
* Any other conditions in addition to the above that the investigators consider may affect study measurements or safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: recruiting 30 patients and 10 controls
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Resting state brain structural measures - white matter and grey matter volumes | 5-7 months post hospital discharge for patients
  Use of MRI sequences to assess grey matter and white matter volume in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Resting state brain structural measures - white matter microstructure | 5-7 months post hospital discharge for patients
  Use of MRI sequences to assess white matter tract distribution in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Resting state cardiac structural integrity - cardiac output | 5-7 months post hospital discharge for patients
  Use of MRI sequences to assess cardiac output at rest in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Resting state cardiac structural integrity - cardiac fibrosis | 5-7 months post hospital discharge for patients
  Use of MRI sequences to look for the degree of fibrosis at rest in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Resting state whole-body fat and muscle volumes | 5-7 months post hospital discharge for patients
  Use of MRI sequence (mDixon) to assess whole-body fat and muscle content in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Resting state myocellular fat content | 5-7 months post hospital discharge for patients
  Use of MR spectroscopy sequence to assess intramyocellular and extramyocellular lipid content in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Dynamic changes in cerebral haemodynamics during low level supine in-bore exercise - cerebral blood flow | 5-7 months post hospital discharge for patients
  MRI sequences will be carried out at rest, during steady-state low level in-bore supine exercise and recovery to assess changes in cerebral blood flow in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Dynamic changes in cerebral haemodynamics during low level supine in-bore exercise - cerebral perfusion | 5-7 months post hospital discharge for patients
  MRI sequences will be carried out at rest, during steady-state low level in-bore supine exercise and recovery to assess changes in cerebral perfusion in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Dynamic changes in cerebral haemodynamics during low level supine in-bore exercise - cerebral oxygen extraction | 5-7 months post hospital discharge for patients
  MRI sequences will be carried out at rest, during steady-state low level in-bore supine exercise and recovery to assess changes in cerebral oxygen extraction in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Dynamic changes in cerebral haemodynamics during low level supine in-bore exercise - cardiac output | 5-7 months post hospital discharge for patients
  MRI sequences will be carried out at rest, during steady-state low level in-bore supine exercise and recovery to assess changes in cardiac output in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Recovery kinetics of skeletal muscle phosphocreatine | 5-7 months post hospital discharge for patients
  Recovery kinetics of phosphocreatine (Pcr) in the gastrocnemius will be measured following its depletion using MR spectroscopy to assess skeletal muscle quality in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Muscle mRNA | 5-7 months post hospital discharge for patients
  Muscle mRNA expression will be determined in skeletal muscle samples obtained from a micro biopsy of the vastus laterals in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Whole body glucose disposal - glucose and insulin concentrations | 5-7 months post hospital discharge for patients
  Oral glucose tolerance test will be used to measure glucose and insulin concentration for whole body glucose disposal in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Whole body glucose disposal - resting energy expenditure | 5-7 months post hospital discharge for patients
  Indirect calorimetry will be used to measure resting energy expenditure for whole body glucose disposal in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.
Motor unit size | 5-7 months post hospital discharge for patients
  Intramuscular electromyography will be used to measure motor unit size in the vastus lateralis in patients with severe Covid-19 at 5-7 months and 11-13 months of discharge from hospital as well as non-Covid, age, gender, BMI and ethnicity matched volunteers.

SECONDARY OUTCOMES:
Clinical and demographic data | 5-7 months post hospital discharge for patients
  age, ethnicity, covid related hospital stay (for patients), covid related interventions (for patients), comorbidities, medications list
muscle strength and function | 5-7 months post hospital discharge for patients
  quadriceps maximum voluntary contraction using cybex dynamometer
hand grip strength | 5-7 months post hospital discharge for patients
  hand grip strength using a hand grip dynamometer will be measured
Short Physical performance battery test (SPPB) | 5-7 months post hospital discharge for patients
  SPPB will be used to assess gait speed, balance and ability to sit up from a chair. Scores within the domains will add up to 4 with 0 being the minimum score
Physical activity | 5-7 months post hospital discharge for patients
  Measuring step count using Sensewear activity arm band
questionnaires for quality of life and symptoms | 5-7 months post hospital discharge for patients
  Fatigue severity score - min score 7 max score 63
questionnaires for quality of life and symptoms | 5-7 months post hospital discharge for patients
  Quality of life as judged by SF-36 - min score 0 max score 100
questionnaires for quality of life and symptoms | 5-7 months post hospital discharge for patients
  Dyspnoea-12 - min score 0 max score 36
questionnaires for quality of life and symptoms | 5-7 months post hospital discharge for patients
  Nottingham activities of daily living - min score 0 max score 22
questionnaires for quality of life and symptoms | 5-7 months post hospital discharge for patients
  Mental health assessed by personal health questionnaire - min score 0 max score 27
questionnaires for quality of life and symptoms | 5-7 months post hospital discharge for patients
  MoCA cognition level - min score 0 max score 30
questionnaires for quality of life and symptoms | 5-7 months post hospital discharge for patients
  Frailty as judged by Rockwood CFS - min score 1 max score 9
blood biomarkers for cardiac function | 5-7 months post hospital discharge for patients
  concentration of troponin
blood biomarkers for cardiac function | 5-7 months post hospital discharge for patients
  concentration of brain natriuretic peptide
blood biomarkers for renal function | 5-7 months post hospital discharge for patients
  calculated glomerular filtration rate
blood biomarkers for liver function | 5-7 months post hospital discharge for patients
  concentration of alanine transaminase
blood biomarkers for skeletal muscle function | 5-7 months post hospital discharge for patients
  concentration of creatine kinase
blood biomarkers for inflammation | 5-7 months post hospital discharge for patients
  concentration of cytokines such as TNF alpha, IL-6 and C-reactive peptide
blood biomarkers for diabetes | 5-7 months post hospital discharge for patients
  Measurement of HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte E Bolton, Prof, Principal Investigator — NIHR Nottingham Biomedical Research Centre, Respiratory theme
Locations (1):
- NIHR Nottingham BRC Respiratory Theme, University of Nottingham and NUH Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Docherty AB, Harrison EM, Green CA, Hardwick HE, Pius R, Norman L, Holden KA, Read JM, Dondelinger F, Carson G, Merson L, Lee J, Plotkin D, Sigfrid L, Halpin S, Jackson C, Gamble C, Horby PW, Nguyen-Van-Tam JS, Ho A, Russell CD, Dunning J, Openshaw PJ, Baillie JK, Semple MG; ISARIC4C investigators. Features of 20 133 UK patients in hospital with covid-19 using the ISARIC WHO Clinical Characterisation Protocol: prospective observational cohort study. BMJ. 2020 May 22;369:m1985. doi: 10.1136/bmj.m1985. PMID 32444460
- [Background] Ronco C, Reis T, Husain-Syed F. Management of acute kidney injury in patients with COVID-19. Lancet Respir Med. 2020 Jul;8(7):738-742. doi: 10.1016/S2213-2600(20)30229-0. Epub 2020 May 14. PMID 32416769
- [Background] Bansal M. Cardiovascular disease and COVID-19. Diabetes Metab Syndr. 2020 May-Jun;14(3):247-250. doi: 10.1016/j.dsx.2020.03.013. Epub 2020 Mar 25. PMID 32247212
- [Background] Narici M, Vito G, Franchi M, Paoli A, Moro T, Marcolin G, Grassi B, Baldassarre G, Zuccarelli L, Biolo G, di Girolamo FG, Fiotti N, Dela F, Greenhaff P, Maganaris C. Impact of sedentarism due to the COVID-19 home confinement on neuromuscular, cardiovascular and metabolic health: Physiological and pathophysiological implications and recommendations for physical and nutritional countermeasures. Eur J Sport Sci. 2021 Apr;21(4):614-635. doi: 10.1080/17461391.2020.1761076. Epub 2020 May 12. PMID 32394816
- [Background] Forster HV, Dempsey JA, Thomson J, Vidruk E, DoPico GA. Estimation of arterial PO2, PCO2, pH, and lactate from arterialized venous blood. J Appl Physiol. 1972 Jan;32(1):134-7. doi: 10.1152/jappl.1972.32.1.134. No abstract available. PMID 5007005
- [Background] Piasecki M, Ireland A, Jones DA, McPhee JS. Age-dependent motor unit remodelling in human limb muscles. Biogerontology. 2016 Jun;17(3):485-96. doi: 10.1007/s10522-015-9627-3. Epub 2015 Dec 14. PMID 26667009
- [Background] Meyerspeer M, Boesch C, Cameron D, Dezortova M, Forbes SC, Heerschap A, Jeneson JAL, Kan HE, Kent J, Layec G, Prompers JJ, Reyngoudt H, Sleigh A, Valkovic L, Kemp GJ; Experts' Working Group on 31P MR Spectroscopy of Skeletal Muscle. 31 P magnetic resonance spectroscopy in skeletal muscle: Experts' consensus recommendations. NMR Biomed. 2020 Feb 10;34(5):e4246. doi: 10.1002/nbm.4246. Online ahead of print. PMID 32037688